CLINICAL TRIAL: NCT03072888
Title: The Effect of Transcutaneous Electrical Nerve Stimulation (TENS) on Pain and Quality of Recovery After Abdominal Hysterectomy
Brief Title: Effects of Transcutaneous Electrical Nerve Stimulation (TENS) Following Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Tuğba Karaman, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TENS
Record Dates: First submitted 2017-02-20; First posted 2017-03-07 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Pain, Acute
Keywords: acute pain; Transcutaneous Electric Nerve Stimulation; Anesthesia Recovery Period
MeSH Terms: conditions — Acute Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS (Experimental): TENS treatment will be apply with 30 minutes sessions seven times per day at the intensity between 9-15 milliamps (mA) which will be adjusted depending on the sensitivity of each individual patient.
  Interventions: Device: TENS
- Control (Sham Comparator): Patients will receive 30 minutes sessions seven times per day of sham TENS therapy without the intensity impulse.
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — Transcutaneous Electrical Nerve Stimulation will be apply
  Other Names: Transcutaneous Electrical Nerve Stimulation

SUMMARY:
The purpose of this study is to evaluate the effect of Transcutaneous Electrical Nerve Stimulation (TENS) in patients after abdominal hysterectomy surgery.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of the Transcutaneous Electrical Nerve Stimulation (TENS) on postoperative pain and quality of recovery in patients following abdominal hysterectomy surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between18-65 undergoing elective abdominal hysterectomy
* ASA (American Society of Anesthesiologist) I,II physical status

Exclusion Criteria:

* Not agreement with the study,Dermatological lesion affecting the electrode place,
* Chronic or preprocedural use of opioids, steroids or psychoactive drugs,
* Allergy to drugs used during trials,
* Previous experience in TENS,
* Kidney, liver, neurological or cardiovascular system disease
* Body mass index>40

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery | At twenty-four hours after surgery
  QoR-40 (Quality of Recovery 40) form will be used for evaluation

SECONDARY OUTCOMES:
Pain | During 24 hours after surgery
  Dynamic and static pain will be evaluated by visual analog scale(VAS)
Analgesic Consumption | During 24 hours after surgery
  Total consumption of analgesic will be recorded
Postoperative Nausea and Vomiting | During 24 hours after surgery
  Nausea and Vomiting scores will be recorded

OTHER OUTCOMES:
Adverse events | During 24 hours after surgery
  The number of adverse events will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa University Medical School, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No